CLINICAL TRIAL: NCT02874378
Title: Effects of Dexmedetomidine on Postoperative Renal Function Recovery After Kidney Transplantation in Adult Patients: Double-Blinded, Randomised Controlled Trial
Brief Title: Effects of Dexmedetomidine on Postoperative Renal Function Recovery After Kidney Transplantation in Adult Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XJTU1AFCT-2016-023
Record Dates: First submitted 2016-08-09; First posted 2016-08-22 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group (Experimental): Dexmedetomidine will be pumped at 0.3μg/kg•h during the operation till 30 minutes before the operation complete. Standard anaesthesia and standard cure are given for all patients.
  Interventions: Drug: Dexmedetomidine
- control group (Placebo Comparator): 0.9%NaCl solution 0.1ml/kg•h during the operation till 30 minutes before the operation complete. Standard anaesthesia and standard cure are given for all patients.
  Interventions: Drug: 0.9%NaCl solution

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Dexmedetomidine Injection
  Arms: study group
Drug: 0.9%NaCl solution
  Other Names: normal saline
  Arms: control group

SUMMARY:
Postoperative renal function recovery is very important to value the operation quality after kidney transplantation. Dexmedetomidine is a selective alpha-2 agonist,enhances urine flow rate and perioperative renal function. Some animal experiments have revealed its beneficial effects against ischemia-reperfusion injury (IRI), our goal is therefore to investigate the effectiveness of a recipient treatment with Dexmedetomidine during operation at reducing Cystatin C level and enhancing renal function after kidney transplantation.

DETAILED DESCRIPTION:
Participants will be randomly assigned, in a 1:1 ratio, to receive Dexmedetomidine or control (0.9 %Sodium Chloride Solution,0.9%NaCl). The randomization sequence will be computer-generated, and randomization will be performed in blocks and will be stratified according to participating center.Dexmedetomidine and 0.9 %NaCl solution will be treated from 10 minutes before anesthesia induction, ending in the last 10 minutes before the operation to complete. Cystatin C level and urine volume (but are not limited to these data) at 1,7,14 days after the transplantation will be recorded. The participation of each patient is scheduled for 14 days.Investigators will research both living and cadaveric kidney transplants.

ELIGIBILITY:
Inclusion Criteria:

Patients underwent renal transplant in the First Affiliated Hospital of Xi'an Jiaotong University.

Exclusion Criteria:

severe comorbidity history: severe cardiac dysfunction, central nervous system disease, endocrine, and history of mental disorders; alcoholic and long-term use of sedatives and opioids history; drug allergy history.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Cystatin C level | 2 weeks

SECONDARY OUTCOMES:
average daily urinary volume | 2 weeks
length of hospital stay (LOS) | an expected average of 2 weeks
Wake up time, extubation time,SAS score,PONV | up to 6 hours
total dosage of remifentanil | up to 4 hours
Cr/GFR improvement | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- the 1st affiliated hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided